CLINICAL TRIAL: NCT05016479
Title: Accelerated rTMS in Gambling Disorder: a Multicentric, Randomized, Sham-controlled Trial
Acronym: arTMSinGD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ITAB - Institute for Advanced Biomedical Technologies (Other)
Responsible Party: Principal Investigator, Mauro Pettorruso, Dr, ITAB - Institute for Advanced Biomedical Technologies
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: richt1ie1
Record Dates: First submitted 2021-08-17; First posted 2021-08-23 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Gambling; Gambling Disorder; Gambling, Pathological; Gambling Problem
Keywords: arTMS; Transcranial Magnetic Stimulation; TMS; Gambling Disorder
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Intervention Model Description: double blind, randomized, sham-controlled with a 1:1 allocation into 2 parallel arms
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: With regard to the treatment, to ensure that both participants and investigators are blind to the condition (active or sham), the selection of the operation mode (15 Hz, sham) will be pre-programmed by member of the that will not be involved in data collection and analysis. Study personnel will not know which mode is being activated. Sham stimulation will use the same coil placement as that used for active stimulation. Outcomes Assessors will not be present during the rTMS sessions.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active arTMS (15 Hz) (Experimental): The treatment involves 15 Repetitive Transcranial Magnetic Stimlation sessions (3/daily for 5 consecutive days, each session lasts 13 min with an interval of 50 min). Coil is placed on the left dorsolateral prefrontal cortex (LDLPFC).The stimulation has a frequency of 15 Hz and a intensity of 120% of the individual resting motor threshold.
  Interventions: Device: Accelerated repetitive Transcranial Magnetic Stimulation
- Sham arTMS (Sham Comparator): Sham group receives the same Repetitive Transcranial Magnetic Stimlation sessions of active compactors. However the interventions in the place group are with a superficial stimulation of scalp muscles only, in order to induce a sensation close to the one experienced with the real rTMS stimulation.
  Interventions: Device: Accelerated repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Accelerated repetitive Transcranial Magnetic Stimulation — arTMS is a non-invasive brain stimulation technique. It will be used a MagPro R30 with a Cool-B80 figure-of-eight coil (MagVenture, Falun, Denmark).
  Other Names: arTMS

SUMMARY:
Background: Gambling disorder (GD), is a behavioral addiction based on keeping play despite medical, economic and social consequences. GD is characterized by progressive and persistent brain circuits alterations (reward, stress, memory, impulse control and cognitive functions), so a possible treatment could be based on neuromodulation of specific brain areas. Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive brain stimulation, which provides magnetic stimuli on certain brain areas parts with short and long-term effects. rTMS has the FDA approval for some neurological (headache) and psychiatric (treatment-resistant depression, obsessive-compulsive disorder) disease. Nowadays several evidence in scientific literature lead to a promise use of rTMS also in addiction field with a possible indication also for GD.

Objectives: the main outcome is to assess symptoms related to GD (craving, play frequencies, money lost) before and after rTMS stimulation on left dorsolateral prefrontal cortex (DLPFC).

Eligibility: Healthy, right-handed adults ages 18-65 with a diagnosis of GD. Design: This is a randomized, sham-controlled study. The study includes two phases:1) a rTMS continued treatment phase and 2) a follow-up without rTMS stimulation (30 days).

In order to be enrolled, participants will be screened with:

* Questionnaires
* Medical history
* Physical exam
* f-MRI

After being enrolled, baseline behavioral and imaging data will be collected. In particular, participants will submit:

* Questionnaires
* Functional MRI
* Cognitive tasks

During the continued rTMS phase, participants with gambling disorder will be randomized to receive real or sham rTMS. RTMS will be delivered during 5 outpatient treatment days, (3 times/die). After the last stimulation and at the end of the 30-days of follow-up period, subjects will undergo the neurocognitive and psychometric evaluation.

Twenty randomized patients of whole enrolled group will undergo fMRI at baseline and at the end of arTMS treatment phase.

Treatment includes:

* rTMS: A weak electrical current passes through a coil placed on the head. During each stimulation day, participants will receive three rTMS sessions (13 min), with a 50 min of interval.
* fMRI: Participants lie on a table that slides into a cylinder that takes pictures of the brain. They respond to images while in the scanner.
* Repeat of screening tests and questionnaires

DETAILED DESCRIPTION:
Repetitive Transcranial Magnetic Stimulation (rTMS) is a neurostimulation technique that consists in the application of magnetic pulses in order to modulate local brain activity, opened up the possibility of interacting with dysfunctional brain circuits, selectively targeting gambling-related cognitive dysfunction.

The main outcome of the present study is to evaluate, in a population of GD patients, the effects of accelerated rTMS (arTMS) applied on Left Dorsolateral Prefrontal Cortex (LDLPFC) in terms of variations in gambling-related symptoms.

In order to investigate the possible effects of arTMS on brain connectivity, a subsample of patients will undergo a functional neuroimaging study based on fMRI.

The study includes 3 psychiatric assessments with psychometric testing: V1 (enrollment), V2 (day 5), V3 (week 4, follow-up).

At Visit 1 (enrollment) the researcher will fully inform the patient about the study, obtaining the patient's informed consent to participate in the study, and will determine the patient's eligibility. Patients will also undergo a battery of cognitive tasks and psychometric evaluation. The same neurocognitive and psychiatric assessment will be repeated during Visit 2 (day 5) and Visit 3 (4 Weeks).

The analysis of the neuroimaging data will allow to evaluate the effect of the active arTMS on brain connectivity (reward system, attention and executive control networks) investigate the association between these evidence and clinical variables.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of Gambling Disorder, based on the Diagnostic and Statistical Manual of Mental Disorder - Fifth Edition (DSM-5);

Exclusion Criteria:

* Current or pre-existing DSM-5 diagnosis of schizophrenia, bipolar disorder, or other psychotic disorder;
* Use in the past 4 weeks of any medication with known pro-convulsant action, including antipsychotic medications, tricyclic antidepressants, and antihistamines drugs;
* Medical history with significant neurological disorder, including organic brain disease, epilepsy, stroke, brain lesions and multiple sclerosis, previous neurosurgery, or personal history of head trauma that resulted in loss of consciousness for > 5 minutes and retrograde amnesia for > 30 minutes;
* Any personal or family history (1st degree relatives) of seizures other than febrile childhood seizures;
* Any psychiatric, medical or social condition whether or not listed above, due to which, according to the judgment of the PI and after any consults if indicated, participation in the study is not in the best interest of the patient;
* For female patients: Pregnancy/breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in gambling behavior assessed by Yale Brown Obsessive Compulsive Scale adapted for Pathological Gambling (PG-YBOCS) | Baseline, after rTMS treatment (5 day), 4 weeks
  To assess the severity of gambling-related symptoms: Yale Brown Obsessive Compulsive Scale adapted for Pathological Gambling (PG-YBOCS), 10-item clinician-administered questionnaire that assess gambling symptoms over a recent time interval
Change in gambling behavior assessed by Gambling Symptom Assessment Scale (G-SAS) | Baseline, after rTMS treatment (5 day), 4 weeks
  a self-rated 5-point Likert scale with total score ranges from 0 to 48
Change in gambling behavior assessed by TimeLine Follow Back (TLFB) - Gambling Version | Baseline, after rTMS treatment (5 day), 4 weeks
  in a multidimension retrospective interview focused on the quantitative assessment of gambling behavior
Change in gambling behavior assessed by Visual Analogue Scale | Baseline, after rTMS treatment (5 day), 4 weeks
  an instrument applied to assess continuum variables, using a horizontal line on which the patient shell point his current state from left vertex (no gambling craving) to right vertex (maximum gambling craving).

SECONDARY OUTCOMES:
Change in attention / hyperactivity symptoms assessed by Adult ADHD Self-Report Scale (ASRS) | Baseline, after rTMS treatment (5 day), 4 weeks
  5-Likert questionnaire to assess the presence of disturbing symptoms attention / hyperactivity
Change in emotional awareness assessed by Toronto Alexithymia Scale (TAS-20) | Baseline, after rTMS treatment (5 day), 4 weeks
  a self-report 5 point Likert scale with 20 items to assess emotional awareness. The total score goes from 20 to 100: non-alexithymia when the score is less than 51, borderline from 51 to 60 and alexithymia if the score is over 60
Change in mood state assessed by Profile of Mood States (POMS) | Baseline, after rTMS treatment (5 day), 4 weeks
  a self-report, 5-point Likert scale to measure the current mood state through six dimensions of affect, including tension-anxiety, depression-dejection, anger-hostility, vigor-activity, fatigue-inertia, and confusion-bewilderment
Change in search for sensations assessed by Sensation Seeking Scale V (SSS-V) | Baseline, after rTMS treatment (5 day), 4 weeks
  a scale created with the purpose of understanding traits as neuroticism, antisocial behavior and psychopathy. There are four different subscales: Thrill and Adventure Seeking, Disinhibition,Experience Seeking, Boredom Susceptibility. Each subscale contains 10 items, making a total of 40 items
Change in hedonic tone assessed by Snaith-Hamilton Pleasure Scale (SHAPS) | Baseline, after rTMS treatment (5 day), 4 weeks
  a 14-item 4-point scale with a total score from 0 to 42
Change in hedonic tone assessed by Temporal Experience of Pleasure Scale (TEPS) | Baseline, after rTMS treatment (5 day), 4 weeks
  a 18-item 6-point scale with a range from 20 to 108
Change in quality of life assessed by Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) | Baseline, after rTMS treatment (5 day), 4 weeks
  to measure the social bonds of the subject with family members, friends, etc; this questionnaire is designed to help assess the degree of enjoyment and satisfaction experienced during the past week. There are 8 subscales : Phisical health, feelings, work, household duties, school/cpurse work, leisure time activities, social relations, general activities.
Change in suicidal behaviours assessed by Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline, after rTMS treatment (5 day), 4 weeks
  The scale identifies specific behaviors which may be indicative of an individual's intent to complete suicide. An individual exhibiting even a single behavior identified by the scale was 8 to 10 times more likely to complete suicide
Change in psychopathological symptoms assessed by SCL-90 | Baseline, after rTMS treatment (5 day), 4 weeks
  measuring both internalizing symptoms (depression, somatization, anxiety) and externalizing ones (aggression, hostility, impulsiveness) of psychiatric patients, general medicine and non-clinical subjects
Change in food craving assessed by Food craving questionnaire (FCI) | Baseline, after rTMS treatment (5 day), 4 weeks
  a self-report 5-point Likert scale assess to evaluate food craving. The questionnaire consists of 28 items collected in 4 subscale: "high fat foods", "sweets", "carbohydrates", "fast foods"
Change in sleep quality assessed by Insomnia severity index (ISI) | Baseline, after rTMS treatment (5 day), 4 weeks
  a self-report 5-point Likert questionnaire to estimate sleep quality in the last month. The total score range is from 0 to 28, in particular: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28)
Change in nicotine craving assessed by Short Tobacco Craving Questionnaire (sTCQ) | Baseline, after rTMS treatment (5 day), 4 weeks
  a Likert based scale (1-7 score) to evaluate nicotine craving. The questionnaire consisted in 4 domines (emotionally, expectancy, compulsivity, purposufullness), each with 3 items
Change in anxiety level assessed by Hamilton Anxiety Scale (HAM-A) | Baseline, after rTMS treatment (5 day), 4 weeks
  a 14-item 5-point scale with a total range score from 0 (min ) to 56 (max), that assesses anxiety symptoms exploring different domains "anxious mood", "tension" or "fears"
Change in depressive symptoms assessed by Hamilton Depression Scale (HAM-D) | Baseline, after rTMS treatment (5 day), 4 weeks
  a interview with 20 items and total score is considered normal with range 0-7
Change in manic symptoms assessed by Young Mania Rating Scale (YMRS) | Baseline, after rTMS treatment (5 day), 4 weeks
  a 11-item interview with total range score form 0 to 60
Change in positive and negative symptoms assessed by Positive Affect and Negative Affect Scales (PANAS) | Baseline, after rTMS treatment (5 day), 4 weeks
  to measure any possible Collateral effect. PANAS is a 20-items 5-poin Likert questionnaire consisted in 2 subscale: Positive Affect Score and Negative Affect Score, with total range from 10 to 50 for each domains
Change in impulsivness assessed by Barratt Impulsiveness Scale (BIS-11) | Baseline, after rTMS treatment (5 day), 4 weeks
  a 11-items self-report questionnaire to evaluate temperamental impulsive traits. BIS-11 consists in 3 subscale: "Attentional Impulsivity", "Motor Impulsivity" and "Nonplanning Impulsivity"
Change in cognitive performance by Iowa gambling task (IGT) | Baseline, after rTMS treatment (5 day), 4 weeks
  a psychological task thought to simulate real-life decision making. Participants are presented with four virtual decks of cards on a computer screen. They are told that each deck holds cards that will either reward or penalize them, using game money. The goal of the game is to win as much money as possible. The decks differ from each other in the balance of reward versus penalty cards
Change in cognitive performance by Go / No-Go Task | Baseline, after rTMS treatment (5 day), 4 weeks
  used to measure a participants capacity for sustained attention and response control. For example, a go/no-go test that requires a participant to perform an action given certain stimuli (e.g., press a button - Go) and inhibit that action under a different set of stimuli (e.g., not press that same button - No-Go).
Change in cognitive performance by Stroop color-word task | Baseline, after rTMS treatment (5 day), 4 weeks
  a neuropsychological test extensively used to assess the ability to inhibit cognitive interference that occurs when the processing of a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute, well-known as the Stroop Effect
Change in cognitive performance by Wisconsin card-sorting task | Baseline, after rTMS treatment (5 day), 4 weeks
  a neuropsychological test of "set-shifting", i.e. the ability to display flexibility in the face of changing schedules of reinforcement. A number of stimulus cards are presented to the participant. The original WCST used paper cards and was carried out with the experimenter on one side of the desk facing the participant on the other

CONTACTS AND LOCATIONS:
Overall Officials: Massimo di Giannantonio, MD, Principal Investigator — ITAB - Institute for Advanced Biomedical

IPD SHARING:
Plan to Share IPD: No